CLINICAL TRIAL: NCT00915005
Title: A Bayesian Randomized Trial of Image-Guided Adaptive Conformal Photon vs Proton Therapy, With Concurrent Chemotherapy, for Locally Advanced Non-Small Cell Lung Carcinoma: Treatment Related Pneumonitis and Locoregional Recurrence
Brief Title: Trial of Image-Guided Adaptive Conformal Photon vs Proton Therapy, With Concurrent Chemotherapy, for Locally Advanced Non-Small Cell Lung Carcinoma: Treatment Related Pneumonitis and Locoregional Recurrence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0133; NCI-2011-01094 (Registry Identifier: NCI CTRP); 2P01CA021239-29A1 (NIH)
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Results first posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: Locally-advanced non-small-cell lung carcinoma; NSCLC; Lung Cancer; Image-Guided Adaptive Conformal Photon; Proton Therapy; Chemotherapy; Treatment Related Pneumonitis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Proton Therapy; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Group 1: Photon Therapy - 74 Gy 37 radiation treatments, given 5 days a week for about 7 1/2 weeks. Each daily treatment should take about 20-30 minutes to complete.
  Paclitaxel 50 mg/m2 by vein 1 time each week for 7 weeks.
  Carboplatin AUC 2 by vein 1 time each week for 7 weeks.
  Interventions: Radiation: Photon Therapy; Drug: Paclitaxel; Drug: Carboplatin
- Group 2 (Experimental): Group 2: Proton Therapy - 74 Gy in 2 CGE per fraction given 5 days a week for about 7 1/2 weeks.
  Paclitaxel 50 mg/m2 by vein 1 time each week for 7 weeks.
  Carboplatin AUC 2 by vein 1 time each week for 7 weeks.
  Interventions: Radiation: Proton Therapy; Drug: Paclitaxel; Drug: Carboplatin
- Group 3 (Experimental): Group 3: Receives either photon or proton therapy, whichever participant's doctor decides is better, for for 6-7 1/2 weeks.
  Paclitaxel 50 mg/m2 by vein 1 time each week for 7 weeks.
  Carboplatin AUC 2 by vein 1 time each week for 7 weeks.
  Interventions: Radiation: Photon Therapy; Radiation: Proton Therapy; Drug: Paclitaxel; Drug: Carboplatin
- Group 4 (Experimental): Photon Therapy - Highest practical dose (74 CGE, 66 CGE) radiation treatments, given 5 days a week for about 7 1/2 weeks. Each daily treatment should take about 20-30 minutes to complete.
  Paclitaxel 50 mg/m2 by vein 1 time each week for 7 weeks.
  Carboplatin AUC 2 by vein 1 time each week for 7 weeks.
  Interventions: Radiation: Photon Therapy; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Radiation: Photon Therapy — Group 1: 74 Gy 37 radiation treatments, given 5 days a week for about 7 1/2 weeks. Each daily treatment should take about 20-30 minutes to complete.
  Arms: Group 1; Group 3; Group 4
Radiation: Proton Therapy — Group 2: 74 Gy in 2 CGE per fraction given 5 days a week for about 7 1/2 weeks.
  Group 3: 66 Gy with conventional fractionation given 5 days a week for about 6-7 1/2 weeks.
  Each daily treatment should take about 20-30 minutes to complete.
  Arms: Group 2; Group 3
Drug: Paclitaxel — 50 mg/m2 by vein 1 time each week for 7 weeks.
  Other Names: Taxol
Drug: Carboplatin — AUC 2 by vein 1 time each week for 7 weeks.
  Other Names: Paraplatin

SUMMARY:
The goal of this clinical research study is to learn if, compared with regular x-ray radiation, proton radiation reduces the risk of developing, treatment-related pneumonitis (TRP) or tumor recurrence (the tumor coming back in the irradiated area after treatment) in patients with lung cancer.

DETAILED DESCRIPTION:
There are 2 types of radiation treatment being used in this study. One type of treatment is proton therapy. Proton therapy is a type of radiation therapy that uses a beam of proton particles (similar to getting an x-ray) to send radiation inside the body to the tumor. The other type of treatment is Image-Guided Adaptive Photon Therapy (IGAPT). IGAPT is a therapy that uses images to help guide the delivery of photon therapy to the tumor. Both of these types of radiation treatment are believed to help doctors to give a full dose of radiation treatment to the tumor while not damaging as much of the healthy tissue around it.

Study Groups If you are found to be eligible to take part in this study, you will go through the standard radiation treatment planning procedure, called the "marking session." After the marking session, a standard photon therapy plan (called Intensity Modulated Radiation Therapy, or IMRT) and a proton plan will be developed. If the radiation oncologist thinks that both the photon and proton plans are acceptable, you will then be randomly assigned to 1 of 2 groups. Participants in Group 1 will receive photon therapy. Participants in Group 2 will receive proton therapy.

The first 20 participants will have an equal chance to be assigned to either group. After at least 20 participants have been enrolled and there has been at least 1 occurrence of pneumonitis and/or tumor recurrence in each treatment Group, the risk of pneumonitis and/or tumor recurrence in all previous participants will be evaluated for each treatment Group, and that information will be used to calculate the chances of being assigned to either Group 1 or Group 2. This calculation will be updated after each occurrence of pneumonitis and/or tumor recurrence and after each participant returns for a follow-up visit. Once these calculations are begun, everyone who joins the study from that point on will be more likely to be assigned to the treatment Group that appears to be better in terms of pneumonitis and/or tumor recurrence.

If the tumor is too large and the standard radiation treatment plan created during the marking session is found not to be acceptable, and the radiation oncologist thinks radiation treatment it is necessary, you will still remain on study and be assigned to a third group. If you are assigned to Group 3, you will receive proton or photon treatment at a lower dose level and/or reduced length of radiation.

If you are assigned to Group 2 and your insurance provider denies reimbursement, you may chose not to receive proton therapy and receive photon therapy instead. If you chose to receive photon therapy, you will be in Group 4.

Radiation Therapy Administration Both radiation therapy treatments (photon and proton) are given through a radiation machine called an accelerator. The radiation therapy administration process is very similar to the way that a CT scan is performed. You will lay on a table and the treatment machine rotates around you without touching your body. Each daily treatment should take about 20-30 minutes to complete. Most of this time is used to position you correctly before the machine is turned on. The actual time used to give the radiation should take about 3-5 minutes each day.

While you are on this study and if you are in Groups 1 or 2, you will receive a total of 37 radiation treatments. Radiation is given 5 days a week for about 7 1/2 weeks.

If you are in Group 1, you will receive photon radiation treatment in the main hospital.

If you are in Group 2, you will receive proton therapy in the proton treatment center (PTC).

If you are in Group 3, you will receive either photon or proton therapy, whichever your doctor decides is better for you, for 6-7 1/2 weeks. If your doctor decides that photon therapy is better you will receive your treatment in the main hospital. If your doctor decides that proton therapy is better you will receive your treatment in the Proton Therapy Center.

If you are in Group 4, you will receive Photon radiation treatment in the main hospital.

Chemotherapy You will receive carboplatin and paclitaxel chemotherapy 1 time a week over 7 weeks. Each treatment will last 3-4 hours. Paclitaxel will be given by vein over 1 hour and carboplatin will be given by vein over 30 minutes. You will receive this chemotherapy combination with radiation therapy, as part of your treatment on this study.

Your chemotherapy may also be decided by your treating medical oncologist as long as the therapy is allowed by the study.

Study Visits During Chemoradiation

At least 1 time each week for all study participants, you will have study tests performed. During this weekly study visit, the following tests and procedures will be performed:

You will have a physical exam. You will be asked about any side effects you may have experienced. Blood (about 2 teaspoons) will be drawn for routine tests.

If the study doctor thinks it is needed, you will have a PET/CT scan performed to check the status of the disease during Week 4 or 5 of treatment.

Length of Study You will remain on study as long you are benefiting. You will be taken off study early if the disease gets worse, you experience intolerable side effects, or your doctor thinks that it is no longer in your best interest to receive the study treatment.

Follow-Up Visits After you have completed chemoradiation, the study staff or study nurse will contact you 1 time each month to ask you about any symptoms you may have until 6 months after chemoradiation. Each phone call should last about 10 minutes.

You will have your first follow-up visit 4-8 weeks after you have completed chemoradiation. You will have additional follow-up visits every 3-4 months for 3 years, every 6 months for the next 2 years, and then 1 time every year after that.

At the first and second follow-up visit the following tests and procedures will be performed:

You will have positron emission tomography (PET)/computed tomography (CT) scans and single proton emission tomography (SPECT) scans to check the status of your lungs and heart if the radiation or medical oncologist thinks it is necessary.

Blood (about 1 teaspoon) will be drawn for routine tests.

If the radiation oncologist or medical oncologist thinks it is needed, at the follow-up visits, you will have breathing function tests performed to check your lung function for up to 1 year after the study treatment is complete. For this test, the radiation oncologist, medical oncologist or study nurse will have you breathe into a special machine. The radiation oncologist or medical oncologist will decide how many tests are to be performed each time.

PET/CT and SPECT scans will be performed again at any time the radiation oncologist or medical oncologist thinks they are needed.

Other tests may be performed if the study doctor (radiation oncologist, medical oncologist, surgeon or pulmonologist) thinks they are needed.

This is an investigational study. Both proton radiotherapy and IGAPT are FDA approved for the treatment of lung cancer.

Up to 250 patients will take part in this multi-center research study. Up to 205 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven, unresected, locoregionally advanced NSCLC without evidence of hematogenous metastases (stage II-IIIB disease according to the 7th edition of the AJCC Staging Manual) with exception as defined by inclusion #2).
2. Patients with solitary brain metastasis without sign of progression in the brain at the time of registration will be eligible for this trial if there is clinical indication for concurrent chemoradiation to the primary disease in the lung.
3. Suitability for concurrent chemoradiation therapy per treating radiation oncologists or treating medical oncologist's: A) Karnofsky performance score of >/= 70, or ECOG 0-1 B) Unintentional weight loss </= 10% during the 3 months before study entry.
4. Receipt of induction chemotherapy followed by referral for concurrent chemoradiation is allowed for this protocol.
5. Measurable disease on chest x-ray, contrast-enhanced CT, or PET scan.
6. Locoregional recurrence after surgical resection, if suitable for definitive concurrent chemoradiation is allowed for this protocol.
7. Forced expiratory volume in the first second (FEV1) >/= 1 liters.
8. Fluorodeoxyglucose (FDG) -PET scan within 3 months before registration. The pretreatment (diagnostic) PET/CT should, whenever possible, be performed together with the 4-D CT simulation. PET images acquired either at the time of simulation or acquired separately should be registered with the planning CT to assist in tumor delineation.
9. Standard pretreatment evaluations (as decided by treating radiation oncologist, medical oncologist, surgeons or pulmonologist), to include MRI or CT scan of the brain, contrast CT scan of the thorax and upper abdomen, Whole-body PET/CT, pulmonary function tests, lung and cardiac single proton emission computed tomography (SPECT), liver function tests (LFT), blood chemistry, renal function tests, and complete blood count.
10. Age >/= 18 years but </= 85 years.
11. A signed specific informed consent form before study entry.

Exclusion Criteria:

1. Small cell histology.
2. Prior thoracic radiotherapy to regions that would result in overlap of radiation therapy fields.
3. Pregnancy (female patients of childbearing potential must practice appropriate contraception).
4. Enrollment in a clinical trial that specifically excludes IGAPT treatment.
5. Body weight exceeds the weight limit of the treatment couch.
6. Oxygen dependent due to preexistent lung disease (COPD, emphysema, lung fibrosis).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhongxing Liao, MD, Study Chair — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Koutroumpakis E, Xu T, Lopez-Mattei J, Pan T, Lu Y, Irizarry-Caro JA, Mohan R, Zhang X, Meng QH, Lin R, Xu T, Deswal A, Liao Z. Coronary artery calcium score on standard of care oncologic CT scans for the prediction of adverse cardiovascular events in patients with non-small cell lung cancer treated with concurrent chemoradiotherapy. Front Cardiovasc Med. 2022 Dec 2;9:1071701. doi: 10.3389/fcvm.2022.1071701. eCollection 2022. PMID 36531700
- [Derived] Cella L, Monti S, Xu T, Liuzzi R, Stanzione A, Durante M, Mohan R, Liao Z, Palma G. Probing thoracic dose patterns associated to pericardial effusion and mortality in patients treated with photons and protons for locally advanced non-small-cell lung cancer. Radiother Oncol. 2021 Jul;160:148-158. doi: 10.1016/j.radonc.2021.04.025. Epub 2021 May 9. PMID 33979653
- [Derived] Gjyshi O, Xu T, Elhammali A, Boyce-Fappiano D, Chun SG, Gandhi S, Lee P, Chen AB, Lin SH, Chang JY, Tsao A, Gay CM, Zhu XR, Zhang X, Heymach JV, Fossella FV, Lu C, Nguyen QN, Liao Z. Toxicity and Survival After Intensity-Modulated Proton Therapy Versus Passive Scattering Proton Therapy for NSCLC. J Thorac Oncol. 2021 Feb;16(2):269-277. doi: 10.1016/j.jtho.2020.10.013. Epub 2020 Oct 22. PMID 33198942
- [Derived] Liao Z, Lee JJ, Komaki R, Gomez DR, O'Reilly MS, Fossella FV, Blumenschein GR Jr, Heymach JV, Vaporciyan AA, Swisher SG, Allen PK, Choi NC, DeLaney TF, Hahn SM, Cox JD, Lu CS, Mohan R. Bayesian Adaptive Randomization Trial of Passive Scattering Proton Therapy and Intensity-Modulated Photon Radiotherapy for Locally Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2018 Jun 20;36(18):1813-1822. doi: 10.1200/JCO.2017.74.0720. Epub 2018 Jan 2. PMID 29293386
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 149 lung non-small cell lung cancer (NSCLC) patients with stage II to IV or recurrent tumor were consented, randomized, and treated under 2008-0133 protocol from June 2009 to March 2014. Intensity-modulated (photon) radiotherapy (IMRT) in 92; passive scattering proton therapy (PSPT) in 57.
Pre-assignment Details: A total of 275 NSCLC patients were consented. 2 patients were consented twice and 1 person denied by Massachusetts General Hospital.47 patients were excluded before the planning process began. 44 patients did not allow random assignment. 32 patients were not treated according to protocol allocation.
Groups:
- Intensity-modulated (Photon) Radiotherapy (IMRT); Passive Scattering Proton Therapy (PSPT): All patients on this trial will receive concurrent weekly carboplatin and paclitaxel chemotherapy with radiation therapy 74 or 66 Gy(RBE).
Period: Overall Study
Arm/Group | Intensity-modulated (Photon) Radiotherapy (IMRT) | Passive Scattering Proton Therapy (PSPT)
Started | 105 | 76
Completed | 92 | 57
Not Completed | 13 | 19
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Patient preferred protons therapy | 6 | 0
Not completed — Insurance denial | 3 | 15

BASELINE CHARACTERISTICS:
Population: There were 149 out of 181 participants randomized, treated and evaluable for data analysis. 32 paticipants off-study (IMRT Arm in 13 and PSPT Arm in 19). Patient- and tumor-related characteristics did not differ between IMRT and PSPT groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensity-modulated (Photon) Radiotherapy (IMRT) | Passive Scattering Proton Therapy (PSPT) | Total
Number analyzed (Participants) | 92 | 57 | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 22 | 61
  >=65 years | 53 | 35 | 88
Age, Continuous [Median (Full Range); unit: years] | 66 [33 to 85] | 67 [39 to 78] | 66.5 [36 to 81.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 24 | 69
  Male | 47 | 33 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 88 | 54 | 142
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 83 | 52 | 135
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 92 | 57 | 149
Karnofsky performance score (KPS) [Number; unit: participants] — The KPS ranking runs from 100 to 0, where 100: "perfect" Normal health, 90: able to carry on normal activity; minor signs or symptoms of disease. 80: normal activity with effort; some signs or symptoms of disease. The KPS was to allow physicians to evaluate a patient's survival. The higher KPS scores, the better treatment outcome.
  participants
    KPS≤ 80 | 61 | 37 | 98
    KPS≥ 90 | 31 | 20 | 51
Smoking history [Number; unit: participants]
  Never | 9 | 3 | 12
  Ever | 83 | 54 | 137
Induction chemotherapy [Number; unit: participants]
  Yes | 61 | 42 | 103
  No | 31 | 15 | 46
Tumor histology [Number; unit: participants]
  Adenocarcinoma | 49 | 30 | 79
  Squamous cell carcinoma | 31 | 17 | 48
  NSCLC unspecified | 7 | 9 | 16
  Large cell | 2 | 1 | 3
  Other | 3 | 0 | 3
Clinical disease stage (American Joint Committee on Cancer [AJCC] 7th Ed) [Number; unit: participants] — American Joint Committee on Cancer [AJCC] 7th Ed:
  Stage IIA: T1-2aN1M0; T2bN0M0 Stage IIB: T2b N1 M0 or T3N0M0 Stage IIIA: T1-2bN2M0 or T3N1-2M0 or T4N0-1M0 Stage IIIB: T1-3N3M0 or T4N2-3M0 Stage IV: M1 The earlier TNM staging, the better treatment outcome
  participants
    AJCC IIA/B | 6 | 8 | 14
    AJCC IIIA | 44 | 21 | 65
    AJCC IIIB | 28 | 24 | 52
    AJCC IV | 5 | 3 | 8
    ACC Recurrence | 9 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: The Incidence and Time to Development of Common Terminology Criteria for Adverse Events, Version 3.0 (CTCAE v3.0) Grade > 3 Treatment-related Pneumonitis (TRP)
Description: The Primary Objective is assess and compare the incidence and time to development of CTCAE v3.0 grade > 3 TRP, among IMRT-Group 1 or PSPT-Group 2 using Bayesian randomization. TRP will be diagnosed clinically by the treating investigator. Any questions regarding the diagnosis or grade of TRP will be resolved by the Protocol PI or by his/her designee(s). The outcomes review committee will meet to discuss each and every patient reported to have developed symptomatic TRP. The final grading of TRP will be decided by the outcomes review committee. Diagnosis of TRP included receipt of radiation that included a certain volume of normal lung, radiographic changes that suggested inflammation consistent with the radiation dose distribution within 12 months after starting chemoradiation, and symptoms attributable to TRP. Final TRP outcomes also were reviewed and approved by independent external experts.
Time Frame: From date of protocol registration until the date of first documented development of CTCAE v3.0 grade > 3 TRP or local failure, whichever occurs first, in both treatment groups, assessed up to 6 years.
Measure: Number; unit: participants
Arm/Group | Intensity-modulated (Photon) Radiotherapy (IMRT) | Passive Scattering Proton Therapy (PSPT)
Number analyzed (Participants) | 92 | 57
participants
  Grade 5 | 2 | 0
  Grade 4 | 0 | 0
  Grade 3 | 6 | 6

2. Primary Outcome: The Incidence and Time to Development of Local Failure (LF)
Description: The Primary Objective is assess and compare the incidence and time to development of local failure, among IMRT-Group 1 or PSPT-Group 2 using Bayesian randomization. Local failure was defined as treatment failure within the planning target volume plus a # 1-cm margin. Images used to report Local failure were registered with radiation dose distribution to accurately assess the location of the failure. Biopsy to confirm Local failure was strongly recommended (Data Supplement). An internal outcomes review committee reviewed each event to ensure objectivity and consistency in reporting Local failure. Final RP outcomes also were reviewed and approved by independent external experts.
  1. Tumor recurrence after achieving complete response,
  2. Residual tumor enlargement of 20% or more on CT according to RECIST criteria,
  3. Recurrence of PET FDG Avidity after achieving complete metabolic response,
  4. Increase in FDG avidity in residual tumor,
  5. Pathologically proven recurrence
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Intensity-modulated (Photon) Radiotherapy (IMRT) | Passive Scattering Proton Therapy (PSPT)
Number analyzed (Participants) | 92 | 57
participants
  Local Failure | 18 | 14
  Local Failure at 12 months | 10 | 6

ADVERSE EVENTS:
Time Frame: From date of protocol registration until the date of documented development of adverse events (AEs) in both treatment groups, assessed up to 6 years.
Arm/Group | Intensity-modulated (Photon) Radiotherapy (IMRT) | Passive Scattering Proton Therapy (PSPT)
All-Cause Mortality (participants affected / at risk) | 2/92 | 0/57
Serious Adverse Events (participants affected / at risk) | 28/92 | 22/57
Other Adverse Events (participants affected / at risk) | 82/92 | 52/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensity-modulated (Photon) Radiotherapy (IMRT) (N=92) | Passive Scattering Proton Therapy (PSPT) (N=57)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (7)
Esophatitis (Gastrointestinal disorders) | 10 (10) | 10 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (8)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 6 (6)
Radiation Induced Dermatitis (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (6)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastro Stricutre (Gastrointestinal disorders) | 2 (2) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Cardiac Ischemia / Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemorrhage, pulmonary/ upper respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dehydration (Gastrointestinal disorders) | 1 (1) | 2 (2)
Fatigue (Congenital, familial and genetic disorders) | 3 (3) | 8 (8)
Fever (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensity-modulated (Photon) Radiotherapy (IMRT) (N=92) | Passive Scattering Proton Therapy (PSPT) (N=57)
Cough (Respiratory, thoracic and mediastinal disorders) | 45 (56) | 28 (32)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 41 (51) | 22 (25)
Esophatitis (Gastrointestinal disorders) | 48 (64) | 37 (45)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 22 (24) | 18 (19)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Radiation Induced Dermatitis (Skin and subcutaneous tissue disorders) | 65 (81) | 45 (57)
Dysphagia (Gastrointestinal disorders) | 35 (38) | 29 (38)
Gastro Stricutre (Gastrointestinal disorders) | 2 (2) | 5 (5)
Odynophagia (Gastrointestinal disorders) | 30 (35) | 18 (23)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 7 (9)
Anorexia (Gastrointestinal disorders) | 28 (31) | 13 (13)
Dehydration (Gastrointestinal disorders) | 7 (7) | 4 (4)
Fatigue (Congenital, familial and genetic disorders) | 67 (91) | 49 (65)
Fever (Congenital, familial and genetic disorders) | 4 (4) | 5 (6)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2013-02-19): https://cdn.clinicaltrials.gov/large-docs/05/NCT00915005/Prot_000.pdf
  • Statistical Analysis Plan (2013-02-19): https://cdn.clinicaltrials.gov/large-docs/05/NCT00915005/SAP_001.pdf